CLINICAL TRIAL: NCT01926379
Title: A Combination Intervention Package for Isoniazid Preventive Therapy in Ethiopia
Brief Title: ENhance Initiation and Retention in Isoniazid Preventive Therapy (IPT) Care for HIV Study (ENRICH Study)
Acronym: ENRICH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AAAK3163; 1R01AI100044-01 (NIH)
Record Dates: First submitted 2013-08-05; First posted 2013-08-20 (Estimated); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: HIV; Tuberculosis
Keywords: Ethiopia; TB; tuberculosis; HIV; IPT; isoniazid; adherence; combination intervention package; retention
MeSH Terms: conditions — Tuberculosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Combination Intervention Package (CIP) (Experimental): Patients who enrolled in HIV care at a CIP site on or after January 1, 2013 and initiate Isoniazid Prevention Therapy (IPT) on or after study initiation on July 1, 2013 will receive the combination intervention components that is a part of the Combination Intervention Package (CIP).
  Interventions: Behavioral: Combination intervention components; Drug: Isoniazid Prevention Therapy
- Standard Of Care (IPT alone) (Other): Patients are screened for tuberculosis (TB) at enrollment in HIV care at a HIV clinic and during each routine clinic visit using a simple symptom questionnaire. Eligible patients will receive the standard of care intervention, Isoniazid Prevention Therapy (IPT), per national guidelines. After IPT initiation, patients return to the HIV clinic monthly for monitoring of side effects, TB symptoms, self-reported 30-day adherence, and to receive a 30-day supply of isoniazid. If adherence problems are noted at any time, the nurse counsels the patient, and if the patient still wants to take IPT, it is continued.
  Interventions: Drug: Isoniazid Prevention Therapy

INTERVENTIONS:
Behavioral: Combination intervention components — The CIP will contain programmatic, structural, and psychosocial components, including:
  1. use of a clinical algorithm by providers;
  2. identification of HIV-infected family members eligible for IPT, using an ICAP-developed family care enrollment form (ICAP - International Center for AIDS Care and Treatment Programs);
  3. review of monitoring data on IPT initiation and adherence during monthly multidisciplinary team meetings;
  4. reimbursement of transportation costs for monthly clinic visits; and
  5. real-time adherence support using IVR via mobile phones and trained Peer Educators.
  Arms: Combination Intervention Package (CIP)
Drug: Isoniazid Prevention Therapy — Standard of care involves Isoniazid Prevention Therapy (IPT) - the administration of Isoniazid (INH) to individuals with latent infection with M. tuberculosis in order to prevent progression to active TB disease.
  Other Names: IPT

SUMMARY:
The purpose of the ENRICH study is to evaluate a combination intervention package (CIP) designed to improve implementation of Isoniazid Preventive Therapy (IPT) among people living with HIV (PLWH) in Ethiopia. The study is a two-arm cluster randomized trial, randomized at the HIV clinic level, which includes 10 HIV clinics in Dire Dawa and Harari, Ethiopia. Clinics are randomized to deliver the combination intervention package (CIP) or standard of care (SOC), with stratification by facility size (<80 or >80 patients enrolled in HIV care per year). The experimental intervention will be delivered to all patients in HIV clinics randomly assigned to CIP who initiated HIV care at the CIP site on or after January 1, 2013 and initiated IPT on or after date of study initiation, July 1, 2013. In HIV clinics assigned to SOC, usual care procedures for provision of IPT will be delivered.

Study Aims and Hypotheses

Aim 1. Characterize and compare the effectiveness of a combination intervention package with standard of care for IPT provision in Ethiopia.

Hypothesis 1.1: IPT initiation for new patients enrolling in HIV care at CIP clinics will be higher than that for newly enrolled patients at SOC clinics.

Hypothesis 1.2: Adherence to and completion of IPT for participants initiating IPT at CIP clinics will be higher than that for those initiating IPT at SOC clinics.

Aim 1a. Assess acceptability of CIP among participants enrolled in HIV care and healthcare providers at CIP clinics. Acceptability will include: 1) perceived barriers and facilitators of uptake and delivery of the intervention package among healthcare providers, and 2) acceptability and utilization of intervention components as well as the overall intervention package among IPT initiators and non-initiators.

Aim 2. Assess the impact of CIP compared with SOC on HIV-related outcomes.

Hypothesis 2: HIV-related outcomes for participants receiving IPT at CIP clinics will be superior to outcomes in participants receiving care at SOC clinics. HIV-related outcomes to be assessed include retention in care and, among those participants receiving antiretroviral therapy (ART), adherence to ART and CD4+ count.

Aim 3. Assess the safety and tolerability of IPT among HIV-infected individuals under routine program conditions in Ethiopia.

Aim 4. Identify patient and program characteristics associated with IPT adherence and completion at SOC sites.

Hypothesis 4.1: IPT adherence and completion will be associated with modifiable patient characteristics, including ART status; knowledge and attitudes about IPT; and social support.

Hypothesis 4.2: IPT adherence and completion will be associated with modifiable program characteristics, including provider/patient ratio, patient tracking, and patient support groups.

DETAILED DESCRIPTION:
The study intervention, combination intervention package (CIP), will contain programmatic, structural and psychosocial components including: 1) health care provider training and mentorship in IPT provision using a clinical algorithm; 2) identification of HIV-infected family members eligible for IPT using a family care enrollment form; 3) review of monitoring data on IPT initiation and adherence during monthly multidisciplinary team meetings; 4) reimbursement of transportation costs to patients for monthly clinic visits; and 5) real-time adherence support using interactive voice response (IVR) via mobile phones and trained peer educators.

Data will be collected from all HIV-infected patients enrolled in HIV care at study sites on or after January 1, 2013; from a subset of patients who initiate IPT and enroll into a measurement cohort (MC); and from program characteristics surveys conducted at the study sites. Routine clinic data from all HIV-infected patients enrolled in HIV care at the 10 participating clinics on or after January 1, 2013 will be used to measure the following outcomes: IPT initiation, completion of IPT, and retention in HIV care. These data will be collected by Research Assistants (RA) by abstracting the following information from the clinic Pre-ART, ART (antiretroviral therapy) and IPT registers during the period of observation on all HIV patients who enrolled in care at a study site on or after January 1, 2013: date of enrollment in HIV care; IPT initiation (yes/no); date of ART initiation (if applicable); IPT outcomes (completion, default, death, stopped, transferred out); TB (tuberculosis) screening results; TB treatment (yes/no); TB treatment outcomes (if applicable); and retention in HIV care.

A measurement cohort of 500 HIV-infected patients initiating IPT on or after July 1, 2013 will be recruited from the 10 clinics (n=250 per study arm). MC participants will be assessed at baseline (enrollment) and monthly intervals for six to nine months, depending on the duration of IPT. Outcomes to be measured among MC participants include: adherence to IPT; adherence to ART (if applicable); change in CD4+ count; and side effects/adverse events. MC participants at both SOC and CIP sites will receive the same assessments. RAs will administer assessments on the day of regularly scheduled clinic visits, including a Baseline interview administered on the day of enrollment (which coincides with the day the participant initiates IPT), monthly follow-up interviews completed throughout IPT, and an end of treatment interview that is completed on the day the participant ends IPT. Participants who miss a study visit will be contacted by study staff and administered the questionnaire over the phone within a 1-week window period of the scheduled clinic visit. RAs will also call the MC participants between clinic visits to conduct unannounced pill counts to assess medication adherence. In addition, 30 MC participants from CIP sites will participate in a qualitative interview to assess feasibility and acceptability of the Interactive Voice Response (IVR) system, one of the interventions in place at CIP sites. Also, three groups will be recruited from CIP clinics to participate in in-depth interviews: IPT initiators, from among participants in the Measurement Cohort (n =15), IPT non-initiators (n=15), and healthcare providers (nurses and peer educators, n=13). In-depth interviews will assess acceptability and preferences of intervention components as well as reasons for IPT non-initiation.

RAs will conduct an assessment of programmatic activities at each HIV clinic prior to study implementation and on a monthly basis thereafter throughout the study period. Clinics in both conditions will receive the same assessments. The RA will administer a brief semi-structured Program Characteristics survey to the ART nurse, who will be most familiar with the day-to-day operations of the HIV clinic. The survey will assess nurse training and mentorship in IPT initiation and HIV treatment; availability and use of an IPT clinical algorithm, IPT and ART adherence training for peer educators (PEs); IPT health education for patients; availability and use of an IPT treatment literacy curriculum, including a flip chart used by PEs; reimbursement for transportation costs for patients; provision of mobile phones, subscriber identification module (SIM) cards and airtime vouchers for HIV patients on IPT; use of IVR messages for medication and appointment reminders and assessment of medication adherence and side effects; and provision of community-based adherence and side effect monitoring by PEs. These data will be used to assess fidelity with the intervention at CIP sites, as well as to measure any potential contamination at SOC sites.

All clinical care will be performed by the clinic staff (nurses and PEs). All study procedures, including participant interviews, pill counts, medical record abstraction, and program characteristics surveys will be performed by study staff (research assistants). Following routine clinic visits, clinic staff will refer patients initiating IPT to study staff, who will screen for eligibility, obtain informed consent, and enroll consenting eligible patients into the MC. In addition, RAs at CIP sites will provide parts of the intervention, including disbursement of mobile phones, SIM cards, airtime vouchers, and cash for transportation reimbursement to eligible patients.

ELIGIBILITY:
Measurement Cohort (MC) Eligibility Criteria

Inclusion Criteria:

* Enrolled in HIV care at a study site on or after 01 January 2013
* Eligible per Ethiopia Federal Ministry of Health guidelines for IPT (without symptoms suggestive of tuberculosis, active hepatitis, regular and heavy alcohol use or peripheral neuropathy) and ready to initiate IPT
* Initiates IPT on or after date of study initiation at any study site
* Aged 18 or older
* Amharic-, Somali-, Oromo/Oromiffa-, Harari- or English-speaking
* Able and willing to provide informed consent within 3 working days of IPT initiation

Exclusion Criteria:

* Children under the age of 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 338 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2016-02 (Actual); Study Completion 2021-05-07 (Actual)

PRIMARY OUTCOMES:
Percentage of patients enrolled in HIV care who initiate IPT | up to 2 years
  IPT initiation is defined as percentage of patients enrolled in HIV care on or after January 1, 2013 who initiate IPT between July 1, 2013 and January 1, 2015. This information will be found through a review of clinic registers.
Percentage of patients who are administered at least 180 doses of IPT within 9 months of IPT initiation | up to 2 years
  IPT completion is defined as at least 180 doses administered within 9 months.

SECONDARY OUTCOMES:
Percentage of participants who attended their most recent HIV clinic appointment 6 months after initiating IPT | up to 2 years
  Retention in HIV care will be measured by percentage of participants who attended their most recent HIV clinic appointment 6 months after initiating IPT.
Percentage of total prescribed ART (antiretroviral therapy) doses ingested for each month of ART treatment for the first 6 months after IPT initiation | up to 2 years
  ART adherence will be measured by percentage of total prescribed ART doses ingested, averaged across medications for each month of treatment, from unannounced pill counts and monthly interviews.
Change in CD4+ count from initiation of IPT to 6 months later | up to 2 years
  Change in CD4 count over 6 months (from initiation of IPT to 6 months later). Routine clinical CD4 test results will be used by study staff and no additional blood draw will be required.
Incidence of adverse events experienced by patients during IPT, as identified through monthly questionnaires and chart review | up to 2 years
  Safety and tolerability will be measured through 1) monthly questionnaires about perceived side effects; and 2) chart review to determine side effects and adverse events requiring discontinuation of isoniazid, as well as cases of TB diagnosed while on IPT.
Percentage of total prescribed IPT doses ingested for each month of IPT treatment | up to 2 years
  IPT adherence will be measured by percentage of total prescribed doses ingested for each month of treatment, from data collected from the unannounced pill counts and monthly interviews.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea A Howard, MD, Principal Investigator — Columbia University
Locations (10):
- Ethiopia (10):
  - Addis Ketema Health Center, Dire Dawa
  - Dire Dawa Health Center, Dire Dawa
  - Gende Gerada Health Center, Dire Dawa
  - Gende Kore Health Center, Dire Dawa
  - Goro Health Center, Dire Dawa
  - Legehare Health Center, Dire Dawa
  - Melka-Jebdu Health Center, Dire Dawa
  - Sabian Health Center, Dire Dawa
  - Arategna Health Center, Harar
  - Jinela Health Center, Harar

IPD SHARING:
Plan to Share IPD: No